CLINICAL TRIAL: NCT01300728
Title: A Randomized Double-Blinded Placebo-Controlled Exploratory Study of Intravenous Immunoglobulin (NewGam 10%) in Amnestic Mild Cognitive Impairment
Brief Title: Study of Intravenous Immunoglobulin in Amnestic Mild Cognitive Impairment
Acronym: MCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Shawn Kile, M.D., MD, Sutter Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVIG-KILE-032010
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Intravenous immunotherapy; Conversion to Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous immunoglobulin (IVIG) (Experimental): IVIG (NewGam 10%)at 0.4 g/kg
  Interventions: Drug: NewGam 10% IVIG
- Saline solution (Placebo Comparator): 0.9% saline solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NewGam 10% IVIG — Subjects will be randomized to receive either an infusion of IVIG at 0.4 g/kg or every 14 days for two months for a total of five infusions.
  Fifty subjects will be enrolled and randomized in a 1:1 IVIG 2.0 g/kg: placebo ratio. Twenty-five subjects will receive IVIG and 25 subjects will receive placebo.
  Arms: intravenous immunoglobulin (IVIG)
Other: Placebo — Subjects will be randomized to receive either an infusion of 0.9% saline solution (placebo) every 14 days for two months for a total of five infusions. Fifty subjects will be enrolled and randomized in a 1:1 IVIG 2.0 g/kg: placebo ratio.
  Arms: Saline solution

SUMMARY:
Patients with mild cognitive impairment (MCI) are a group recognized at being at high risk of progressing to Alzheimer disease. Treatment of MCI with immunotherapy with intravenous immunoglobulins (IVIG) could potentially reduce the risk of progression to Alzheimer disease.

This study will evaluate the efficacy of intravenous immunoglobulin in patients with MCI over 24 months after the first infusion. This study will also document conversion from MCI to Alzheimer's Disease.

DETAILED DESCRIPTION:
Screening procedures at visit 1 will take place up to 28 days prior to Visit 2 (Day 1) dosing. Screening labs and assessments will be performed during the screening period. A brain MRI will be obtained as standard of care within 6 months prior to the screening period. The first dose of study drug is administered on Day 1. Visits 2 through 6 have a ±1 day window and occur every 14 days over two months. The investigator will determine if a subject is suitable to continue following the missed infusion. Visits 7 through 12 (Month 4 through Month 24) have a ±7 day window.

All study screening data from Visit 1 including laboratory results must be reviewed for study eligibility prior to receiving first dose of study drug. Visit 2 physical exams and neurological exams prior to infusion may occur within 72 hours prior to the first infusion. Prior to infusion, a review of concomitant medications and adverse events takes place to ensure that no excluded medications have been added or medication discontinued or dose changed that were required to have been stable. If the subject continues to be eligible for enrollment, the subject will be randomized, infused with study medication and will remain in the infusion clinic for at least 4 hours following the start of the infusion for safety assessments on Visit 2 (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 50 to < 85 years old.
2. Diagnosis of Mild Cognitive Impairment, Amnestic type (single or multi domain) according to Petersen criteria (Appendix B) and supported by a CDR score of 0.5.
3. Mini-Mental State Examination (MMSE) score of 24-30, inclusive.
4. Rosen Modified Hachinski Ischemic score ≤ 4.
5. Willing to consent to Apolipoprotein E (ApoE) testing and agree to disclose Apolipoprotein E4 (ApoE4) status. Previous ApoE testing will be accepted.
6. Receiving stable doses of medication(s) for the treatment of non-excluded medical condition(s) for at least 30 days prior to screening.
7. Ability to attend all clinical visits and have an informant capable of accompanying the subject on specific clinic visits for two years or the duration of the study.
8. The subject's collaborative informant (support person) must be someone who has known the subject for at least 4 years; agrees to have at least 2 separate communications with the study participant per month for the duration of the study (one of these communications must be in person); and attends and completes the CDR interview at 8 study visits along with the subject.
9. Fluency in English and evidence of adequate premorbid intellectual functioning.
10. Adequate manual dexterity, visual, and auditory abilities to perform all aspects of the cognitive and functional assessments.
11. Venous access suitable for repeated infusion and phlebotomy.

Exclusion criteria:

1. Has significant neurological disease, other than a-MCI that may affect cognition.
2. History of clinically evident stroke or history of clinically significant carotid or vertebrobasilar stenosis or plaque.
3. History of seizures, excluding febrile seizures in childhood.
4. Brain MRI shows moderate or severe cortical or hippocampal atrophy.
5. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, CSF shunts, claustrophobia, metal fragments or foreign objects in the eyes, skin, or body that would contraindicate a brain MRI scan.
6. Current presence of a clinically significant major psychiatric disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR).
7. History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma, and squamous cell carcinoma of the skin.
8. Uncontrolled hypertension (diastolic BP> 100 mmHg or systolic BP> 160 mmHg, sitting).
9. History or evidence of any clinically significant autoimmune disease or disorder of the immune system (eg., Crohn's Disease, Rheumatoid Arthritis)
10. Women of childbearing potential.
11. Weight greater than 120 kg (264 lbs).
12. Excessive smoking defined as more than 20 cigarettes per day.
13. History of alcohol or drug dependence or abuse as defined by DSM-IV criteria within the last 2 years.
14. Severe liver or kidney disease verified by the PI review of alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine.
15. Known coagulopathy, thrombosis, or low platelet count.
16. Known deficiency to Immunoglobulin A (IgA).
17. Positive serology for Hepatitis B or C, or HIV.
18. Concurrent or prior treatment with cholinesterase inhibitors and/or memantine, or Axona for cognitive enhancement. Exceptions (e.g. brief exposure to one of these medications) may be authorized if agreed upon by PI and sub-I.
19. Concurrent use of anticholinergic drugs including diphenhydramine.
20. Current use of anticonvulsant drugs for seizures, antiparkinson drugs, anticoagulant medications (except the use of aspirin 325 mg/day or less, plavix, aggrenox, and persantine but not for stroke).
21. Concurrent use of opioid pain relievers and related synthetic derivatives.
22. Use of experimental medications for AD or any other investigational medications or devices within 60 days prior to screening or within 5 half-lives of use of such a medication prior to screening, whichever is longer.
23. Prior treatment with IVIG or other experimental immunotherapeutic or vaccine for MCI or AD, or prior treatment with a biological product for the treatment of a-MCI or AD.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Kile, M.D., Principal Investigator — Sutter Health
Locations (1):
- Sutter Neuroscience Medical Group, Sacramento, California, United States

REFERENCES:
- [Background] Relkin NR, Szabo P, Adamiak B, Burgut T, Monthe C, Lent RW, Younkin S, Younkin L, Schiff R, Weksler ME. 18-Month study of intravenous immunoglobulin for treatment of mild Alzheimer disease. Neurobiol Aging. 2009 Nov;30(11):1728-36. doi: 10.1016/j.neurobiolaging.2007.12.021. Epub 2008 Feb 21. PMID 18294736
- [Result] Kile S, Au W, Parise C, Rose K, Donnel T, Hankins A, Chan M, Ghassemi A. IVIG treatment of mild cognitive impairment due to Alzheimer's disease: a randomised double-blinded exploratory study of the effect on brain atrophy, cognition and conversion to dementia. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):106-112. doi: 10.1136/jnnp-2015-311486. Epub 2015 Sep 29. PMID 26420886
- [Derived] Kile S, Au W, Parise C, Rose K, Donnel T, Hankins A, Au Y, Chan M, Ghassemi A. Five-year outcomes after IVIG for mild cognitive impairment due to alzheimer disease. BMC Neurosci. 2021 Aug 6;22(1):49. doi: 10.1186/s12868-021-00651-2. PMID 34362303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-two participants were randomized; however, 2 participants in the IVIG group did not complete the series of 5 infusions, and 1 placebo participant was excluded due to significant language symptoms which were a barrier to cognitive testing. This resulted having a data set consisting of a total of 49 subjects.
Groups:
- Intravenous Immunoglobulin (IVIG): IVIG (NewGam 10%)at 0.4 g/kg
  NewGam 10% IVIG: Subjects will be randomized to receive either an infusion of IVIG at 0.4 g/kg or every 14 days for two months for a total of five infusions.
  Fifty subjects will be enrolled and randomized in a 1:1 IVIG 2.0 g/kg: placebo ratio. Twenty-five subjects will receive IVIG and 25 subjects will receive placebo.
Period: Overall Study
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Started | 26 | 26
Completed | 24 | 25
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.26 (7.91) | 72.40 (7.36) | 72.32 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mean Cognitive Performance [Mean (Standard Deviation); unit: units on a scale] — 12 month cognitive performance in treatment (IVIG/placebo) is measured by:
  * Alzheimer Disease Assessment Scale-cognitive subscale (ADAS-cog)
    * Scale from 0 to 85 (0 is best cognitive performance)
    * Score is the sum of 12 sub-scales.
  * Mini Mental State Exam (MMSE)
    * Scale from 0 to 30 (30 is best cognitive performance)
    * Score is the sum of 11 sub-scales.
  * Clinical Dementia Rating - Sum of Boxes (CDR-SB)
    * Scale is 0 to 18 (0 is best cognitive performance)
    * Score is the sum of 6 sub-scales
  units on a scale
    MMSE | 26.75 (2.15) | 26.44 (2.6) | 26.59 (2.37)
    ADAS-cog | 10.63 (4.23) | 10.29 (5.68) | 10.46 (4.97)
    CDR_SB | 1.96 (0.95) | 1.58 (0.90) | 1.78 (0.94)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Percent Change in Ventricular Volume (APCV) as Measured by MRI
Description: Change in ventricular volumetric as measured by MRI at baseline, 12, and 24 months following the first infusion of either 0.4 g/kg NewGam or 0.9% saline solution(placebo) every 14 days x 5.
  Participants will also be classified as early MCI (EMCI) if baseline CDR-SB is less than 1.5, and late MCI (LMCI) if CDR-SB is greater than or equal to 1.5.
Time Frame: Baseline, 12, and 24 month MRI evaluation
Population: Annualized Percent Change in ventricular volume (APCV) at 12 and 24 months was computed as:
  ((12 or 24 month volume) - (Baseline volume))/(Baseline volume)/(Time (years) between Baseline and 12 or 24 month visit)
Measure: Mean (Standard Deviation); unit: percent change per participant year
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Number analyzed (Participants) | 24 | 25
percent change per participant year
  APCV Baseline to12 months | 5.87 (3.91) | 8.14 (4.43)
  APCV Baseline to 24 months | 6.26 (4.17) | 7.08 (4.05)

2. Secondary Outcome: Number of Participants Who Converted From Amnestic Mild Cognitive Impairment (a-MCI) to Alzheimer Disease (AD)
Description: The National Institute of Neurological and Communicative Disorders and Stroke - Alzheimers Disease and Related Disorders Association (NINCDS-ADRDA) Alzheimer's Criteria were proposed in 1984 by NINCDS-ADRDA criteria for diagnosing Alzheimer Disease and Clinical Dementia Rating (CDR) will be used to determine conversion from a-MCI to AD.
Time Frame: Baseline to 24 months
Measure: Number; unit: participants
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Number analyzed (Participants) | 24 | 25
participants | 16 | 10

3. Secondary Outcome: Change in Ventricular Volume in Patients With Positive Cerebrospinal Fluid (CSF) Aβ1-42/CSF P-Tau181P Alzheimer Signature
Description: Mean ventricular volume (cubic centimeters) in patients with positive cerebrospinal fluid (CSF) Aβ1-42/CSF P-Tau181P Alzheimer signature at 24 months following infusion
Time Frame: Baseline to 24 months following infusion
Measure: Mean (Standard Deviation); unit: cubic centimeters (cc)
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Number analyzed (Participants) | 16 | 15
cubic centimeters (cc)
  Aβ42 (cc) | 294.00 (96.55) | 353.41 (112.99)
  tau (cc) | 107.47 (58.65) | 96.18 (65.47)
  p-tau (cc) | 43.59 (19.90) | 39.47 (30.27)

4. Secondary Outcome: Mean Cognitive Performance at 12 Months
Description: 12 month cognitive performance in treatment (IVIG/placebo) is measured by:
  * Alzheimer Disease Assessment Scale-cognitive subscale (ADAS-cog)
    * Scale from 0 to 85 (0 is best cognitive performance)
    * Score is the sum of 12 sub-scales.
  * Mini Mental State Exam (MMSE)
    * Scale from 0 to 30 (30 is best cognitive performance)
    * Score is the sum of 11 sub-scales.
  * Clinical Dementia Rating - Sum of Boxes (CDR-SB)
    * Scale is 0 to 18 (0 is best cognitive performance)
    * Score is the sum of 6 sub-scales
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Number analyzed (Participants) | 24 | 25
units on a scale
  Mini Mental State Exam (MMSE) | 26.04 (3.76) | 25.38 (4.28)
  Alzheimer's Disease Assessment Scale (ADAS-Cog) | 11.03 (6.66) | 11.00 (9.14)
  Clinical Dementia Rating Sum of Boxes (CDR-SB) | 2.7 (1.63) | 2.65 (2.13)

5. Secondary Outcome: Mean Cognitive Performance at 24 Months
Description: 24 month cognitive performance in treatment (IVIG/placebo) is measured by:
  * Alzheimer Disease Assessment Scale-cognitive subscale (ADAS-cog)
    * Scale from 0 to 85 (0 is best cognitive performance)
    * Score is the sum of 12 sub-scales.
  * Mini Mental State Exam (MMSE)
    * Scale from 0 to 30 (30 is best cognitive performance)
    * Score is the sum of 11 sub-scales.
  * Clinical Dementia Rating - Sum of Boxes (CDR-SB)
    * Scale is 0 to 18 (0 is best cognitive performance)
    * Score is the sum of 6 sub-scales
Time Frame: 24 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
Number analyzed (Participants) | 24 | 25
units on a scale
  Mini Mental State Exam (MMSE) | 24.00 (4.91) | 24.46 (4.79)
  Alzheimer's Disease Assessment Scale (ADAS-Cog) | 15.39 (10.55) | 13.25 (11.77)
  Clinical Dementia Rating Sum of Boxes (CDR-SB) | 4.33 (3.48) | 3.37 (2.73)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Intravenous Immunoglobulin (IVIG) | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/24 | 2/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 1/24 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Immunoglobulin (IVIG) (N=24) | Saline Solution (N=25)
Insomnia (General disorders) | 1 (1) | 0 (0) — Severity = mild
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severity = mild
Low grade fever (General disorders) | 1 (1) | 0 (0) — Severity = mild
Headache (General disorders) | 1 (1) | 0 (0) — Severity = moderate
Chills (General disorders) | 0 (0) | 1 (1) — Severity = moderate
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Severity = mild
Fatigue (General disorders) | 0 (0) | 1 (1) — Severity = mild
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) — Severity = mild
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Severity = mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT01300728/Prot_SAP_000.pdf